CLINICAL TRIAL: NCT02851472
Title: Prevention of Transfusion Related Acute Gut Injury (TRAGI) in Extremely Low Gestational Age Neonates (ELGAN) Neonates Using iNO
Brief Title: Prevention of Transfusion Related Acute Gut Injury (TRAGI) in Extremely Low Gestational Age Neonates (ELGANs) Using iNO
Acronym: iNO-TRAGI
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: New York Medical College (Other)
Collaborators: Stony Brook University (Other); Baystate Medical Center (Other); East Carolina University (Other); New York University (Other)
Responsible Party: Principal Investigator, Edmund LaGamma, Chief of Neonatology, New York Medical College
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: FDA IND 126254
Record Dates: First submitted 2016-07-20; First posted 2016-08-01 (Estimated); Last update posted 2019-04-24 (Actual); Status verified 2019-04

CONDITIONS: Anemia
Keywords: TRAGI (transfusion related acute gut injury); inhaled nitric oxide (iNO); prematurity; PRBC transfusion; NEC (necrotizing enterocolitis); NIRS (near infrared spectroscopy); ELGAN (extremely low gestational age neonate)
MeSH Terms: conditions — Anemia; Premature Birth; Enterocolitis, Necrotizing

STUDY DESIGN:
Intervention Model Description: subjects are randomize into either of two groups: intervention or placebo
Who Masked: Participant, Care Provider, Investigator
Masking Description: iNO vs nitrogen will be administered from tanks labeled with a code number that is known by the manufacturer and a campus safety officer but masked to investigators and to bedside personnel.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Inhaled Nitric Oxide (Experimental): iNO will be given at 20 ppm, continuous, via inhalation before (1 hour), during (3 hours) and after (2 hours) elective blood transfusion and NIRS monitoring
  Interventions: Drug: Inhaled Nitric Oxide
- Placebo (Active Comparator): Placebo gas (nitrogen) will be given continuous, via inhalation at the same ppm, before (1 hour), during (3 hours) and after (2 hours) elective blood transfusion and NIRS monitoring
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Inhaled Nitric Oxide — Nitric oxide gas will be added to the inhaled gas mixture that the patient was already receiving at baseline, using standard of care gas delivery systems adapted specifically for this study.
  Other Names: iNO
  Arms: Inhaled Nitric Oxide
Drug: Placebo — Placebo gas (nitrogen) will be added to the inhaled gas mixture that the patient was already receiving at baseline, using standard of care gas delivery systems specifically adapted for this study.
  Other Names: Control
  Arms: Placebo

SUMMARY:
The investigators seek to determine whether providing inhaled nitric oxide (iNO; a vasodilator) will improve the delivery of oxygen to the brain, kidney and intestines of preterm neonates during and after the subject receives a packed red blood cell transfusion (PRBC) for anemia vs. baseline period. The investigators will observe the effect of inhaled nitric oxide vs. placebo at these body sites to determine whether iNO will alter the fractional tissue oxygen extraction. Treatment and control groups will be compared to each other at equivalent epochs as will individual patients before, during and after the PRBC transfusion.

DETAILED DESCRIPTION:
Selection criteria: 1) Neonates 24 0/7 to 27 6/7 weeks gestational age (GA) 2) More than 2 weeks postnatal age. 3) Anemia with Hct less than 28 % 4) >50 % total daily fluids is enteral 5) History of at least 1 prior PRBC transfusion ELGANs admitted to the neonatal intensive care unit (NICU) will be screened for the study. If patients meet the selection criteria, parents will be approached to obtain informed consent. Then the patient will be randomized to either iNO or placebo group before treatment. The treating physician will make the decision regarding timing of the PRBC transfusion to treat anemia for the subject.

During the period of observation, near infrared spectroscopy (NIRS) monitoring will be performed on all enrolled subjects during which a non-invasive probe will be attached to the skin at 3 sites simultaneously- on abdomen below umbilicus, flank/back, and forehead for calculation of fractional tissue oxygen extraction ( FTOE) in conjunction with concurrent pulse oximetry recordings.

Conventional vital signs, blood gas, lactate, haptoglobin and cytokines will be measured before and after the PRBC transfusion

ELIGIBILITY:
Inclusion Criteria:

* Neonates 24 0/7 to 27 6/7 weeks gestational age
* More than 2 weeks postnatal age.
* Anemia with hematocrit (Hct) less than 28 %
* More than 50 % total daily fluids is enteral
* History of at least 1 prior PRBC transfusion (preferably same donor)

Exclusion Criteria:

* Prior history of necrotizing enterocolitis (NEC) to avoid a confounder
* Clinically significant patent ductus arteriosus (PDA) requiring treatment (Rx) within 24h
* Hypotensive for age or active bleeding
* < 50% of total fluids are enteral (breast milk or formula)
* Major congenital or surgical malformations
* Known chromosomal anomalies detected by antepartum testing or direct physical examination with subsequent postnatal laboratory confirmation
* Absence of parental or treating physician consent
* A concurrent randomized clinical trial (RCT) with another randomized drug
* Death expected < 48h
* Another major concern by the treating physician that either mandates or prohibits study treatment such as known adverse reaction to prior transfusion (Tx)

Min Age: 2 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2019-02-06 (Actual); Primary Completion 2021-02-05 (Estimated); Study Completion 2021-06-30 (Estimated)

PRIMARY OUTCOMES:
Increased NIRS oxygenation after a PRBC transfusion in iNO treated neonates vs Placebo | 19 hours
  The investigators hypothesize that NIRS signal will be significantly higher in the iNO treated group during the 2nd hour after transfusion is concluded vs Placebo. NIRS will be measured continuously and averaged every 5 minutes to create a single hourly point for each subject before and after the transfusion for statistical analysis.

SECONDARY OUTCOMES:
Lower fractional tissue oxygen extraction (FTOE) in iNO treated neonates after PRBC transfusion vs Placebo | 19 hours
  FTOE will be calculated from the 5 minute epochs of the recorded pulse oximeter and NIRS devices. The investigators hypothesize that FTOE will be significantly lower (i.e. improved) in the iNO treated group during the 2nd hour after transfusion is concluded vs Placebo. One entire hour before and another after the transfusion will be combined for each patient for statistical analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Edmund LaGamma, MD, Principal Investigator — New York Medical College
Locations (4):
- United States (4):
  - Baystate Children's Hospital, Springfield, Massachusetts
  - Stony Brook Children's Hospital, Stony Brook, New York
  - Maria Fareri Childrens Hospital, Valhalla, New York
  - East Carolina University, Greenville, North Carolina

IPD SHARING:
Plan to Share IPD: Yes
After publication of the primary manuscript.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: After publication of the primary manuscript
Access Criteria: Data available if there is a well thought-out plan from a credible investigator who is exeprineced in neonatology, transfusion medicine or control of the microcirculation via nitric oxide.

REFERENCES:
- [Result] La Gamma EF, Blau J. Transfusion-related acute gut injury: feeding, flora, flow, and barrier defense. Semin Perinatol. 2012 Aug;36(4):294-305. doi: 10.1053/j.semperi.2012.04.011. PMID 22818551
- [Result] Mintzer JP, Parvez B, Chelala M, Alpan G, LaGamma EF. Monitoring regional tissue oxygen extraction in neonates <1250 g helps identify transfusion thresholds independent of hematocrit. J Neonatal Perinatal Med. 2014 Jan 1;7(2):89-100. doi: 10.3233/NPM-1477213. PMID 25104129
- [Result] Mintzer JP, Parvez B, La Gamma EF. Regional Tissue Oxygen Extraction and Severity of Anemia in Very Low Birth Weight Neonates: A Pilot NIRS Analysis. Am J Perinatol. 2018 Dec;35(14):1411-1418. doi: 10.1055/s-0038-1660458. Epub 2018 Jun 15. PMID 29906796
- [Result] Mintzer JP, Parvez B, Alpan G, LaGamma EF. Effects of sodium bicarbonate correction of metabolic acidosis on regional tissue oxygenation in very low birth weight neonates. J Perinatol. 2015 Aug;35(8):601-6. doi: 10.1038/jp.2015.37. Epub 2015 Apr 30. PMID 25927273
- [Result] Mintzer JP, Parvez B, La Gamma EF. Umbilical Arterial Blood Sampling Alters Cerebral Tissue Oxygenation in Very Low Birth Weight Neonates. J Pediatr. 2015 Nov;167(5):1013-7. doi: 10.1016/j.jpeds.2015.08.016. Epub 2015 Sep 1. PMID 26340878
- [Result] LaGamma, EF, Feldman, A, Mintzer, J, Lakshminrusimha, S, Alpan, G. Red Blood Cell Storage in Transfusion-Related Acute Gut Injury. NeoReviews 16 (7): e420-e430, 2015